CLINICAL TRIAL: NCT02775552
Title: Impact Evaluation of Alive & Thrive's Multi-Sectoral Community-Based Approach to Improving Infant and Young Child Feeding in Amhara, Ethiopia
Brief Title: Impact Evaluation of a Multi-Sectoral Community-Based Approach to Improving Infant and Young Child Feeding in Amhara, Ethiopia
Acronym: A&T-2 Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: FHI 360 (Other); Save the Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 601011
Record Dates: First submitted 2016-05-12; First posted 2016-05-17 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Exclusive Breastfeeding; Complementary Feeding
Keywords: Child Nutrition; Breastfeeding; Complementary Feeding; Infant and Young Child Feeding; Social and Behavior Change Communication; Ethiopia
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A&T intervention areas (Experimental)
  Interventions: Behavioral: A&T community-based interventions; Behavioral: Mass media
- Comparison areas (Active Comparator): (Receive standard government services)
  Interventions: Behavioral: Mass media

INTERVENTIONS:
Behavioral: A&T community-based interventions — 1. Interpersonal communication delivered by health workers and community volunteers at the health post and during home visits to:
     - Increase mothers' knowledge about adequate child feeding practices
  2. Interpersonal communication delivered by agricultural extension workers to:
     - Increase fathers' knowledge about nutrition-sensitive agriculture and child feeding
  3. Community mobilization activities to:
     * Raise awareness of child feeding practices among community members, and increase support to mothers (enhanced community conversations)
     * Increase mothers' knowledge about preparation of complementary foods (cooking demonstrations)
     * Raise awareness of adequate child feeding during fasting among family and community members (church sermons)
  4. Enhanced training of government health and agricultural extension workers in infant and young child feeding to:
     * Improve their ability to provide timely and appropriate information and support to mothers and families
  Arms: A&T intervention areas
Behavioral: Mass media — Radio campaign - radio drama series, spots, and jingles

SUMMARY:
Alive & Thrive is an initiative that aims to scale up nutrition to save lives, prevent illness, and ensure healthy growth and development through improved infant young child feeding (IYCF) practices. The purpose of this study is to evaluate whether the Alive & Thrive intervention package, consisting of interpersonal communication, community mobilization activities, and radio campaign, can increase complementary feeding practices (minimum dietary diversity and minimum meal frequency) while sustaining exclusive breastfeeding rate among children less than two years of age. The impact evaluation uses a cluster-randomized design where 20 geographic clusters (woredas/districts) were randomized to two study arms - 10 intervention areas and 10 comparison areas. Repeated cross-sectional baseline and endline surveys will be used to assess program impact.

DETAILED DESCRIPTION:
In Amhara, the median duration of exclusive breastfeeding (4.6 months) is the highest among all the other regions in the country, but complementary feeding indicators lag behind (2% minimum dietary diversity and 34% minimum meal frequency). As a result, A&T's program emphasis will be placed on increasing mothers' knowledge and skills to improve complementary feeding practices without compromising exclusive breastfeeding. Given the short duration of implementation, the goal is to show that it is possible to achieve behavior change related to IYCF through a multi-sector approach. The purpose of this study is to evaluate whether the Alive & Thrive intervention package, consisting of interpersonal communication, community mobilization activities, and radio campaign, can increase select complementary feeding practices (minimum dietary diversity and minimum meal frequency increased by 10 percentage points) while sustaining exclusive breastfeeding rate among children less than two years of age.

A cluster randomized design with repeated cross-sectional surveys at baseline (2015) and endline (2017) is used to assess impact of the A&T interventions in three western zones of Amhara, Ethiopia. In the three zones, 20 woredas (districts) were randomly assigned as 10 intervention and 10 comparison/control areas. A&T intervention areas are expected to receive intensive IYCF social and behavior change communication activities as well as exposure to a region-wide radio campaign. In accordance with program objectives, sample sizes for the household survey were estimated to detect changes in the three main impact indicators - sustained exclusive breastfeeding, improved minimum dietary diversity, and improved minimum meal frequency. The estimated household sample sizes are 400 children 0-5.9 months old for exclusive breastfeeding in the A&T intervention areas only and 1350 children 6-23.9 months old per study arm for complementary feeding practices, for a total sample size of 3100 children 0-23.9 months of age. Infant feeding practices will be assessed using before- and after- intervention-comparison area group differences between the baseline survey (March-April 2015) and endline survey (March-April 2017). In addition, surveys of frontline workers will help document their awareness and knowledge about IYCF, training, supervision, and delivery of interventions to beneficiary households.

ELIGIBILITY:
Inclusion Criteria:

* Gives informed consent
* Being aged from 15 to 49 years (women of reproductive age)
* Has at least one infant less than 24 months old who is currently alive and lives with her

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3120 (Actual)
Dates: Start 2015-03; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Exclusive breastfeeding among children aged 0-5.9 months in the intervention areas only | 2 years after baseline in a cross-sectional endline survey scheduled for March-April 2017
  The proportion of infants aged less than 6 months who were exclusively breastfed on the day preceding the interview.
Minimum dietary diversity among children aged 6-23.9 months | 2 years after baseline in a cross-sectional endline survey scheduled for March-April 2017
  The proportion of children aged 6-23.9 months months who received foods from 4 or more food groups on the day preceding the interview.
Minimum meal frequency of (semi) solid or soft foods among children aged 6-23.9 months | 2 years after baseline in a cross-sectional endline survey scheduled for March-April 2017
  The proportion of children aged 6-23.9 months who received (semi) solid or soft foods the minimum number of times or more on the day preceding the interview.

SECONDARY OUTCOMES:
Early initiation of breastfeeding among children aged 0-5.9 months in the intervention areas only and among children aged 6-23.9 months in intervention and comparison areas | 2 years after baseline in a cross-sectional endline survey scheduled for March-April 2017
  The proportion of children aged less than 24 months who were breastfed within 1 hour of birth.
Continued breastfeeding at 1 year among children aged 12-15.9 months | 2 years after baseline in a cross-sectional endline survey scheduled for March-April 2017
  The proportion of children aged 12-15.9 months who were breastfed on the day preceding the interview.
Timely introduction of (semi) solid or soft foods among children aged 6-8.9 months | 2 years after baseline in a cross-sectional endline survey scheduled for March-April 2017
  The proportion of infants aged 6-8.9 months who received (semi) solid or soft foods on the day preceding the interview.
Minimum acceptable diet among children aged 6-23.9 months | 2 years after baseline in a cross-sectional endline survey scheduled for March-April 2017
  The proportion of children aged 6-23.9 months who received a minimum acceptable diet (minimum dietary diversity and minimum meal frequency) on the day preceding the interview.
Consumption of iron-rich foods among children aged 6-23.9 months | 2 years after baseline in a cross-sectional endline survey scheduled for March-April 2017
  The proportion of children aged 6-23.9 months who received an iron-rich or iron-fortified food on the day preceding the interview.
Mother's accurate knowledge of adequate child feeding practices | 2 years after baseline in a cross-sectional endline survey scheduled for March-April 2017
  Proportion of mothers who report correct knowledge about breastfeeding and complementary feeding practices based on questionnaire
Mother's beliefs, self-efficacy, and perceptions of social norms about child feeding during fasting | 2 years after baseline in a cross-sectional endline survey scheduled for March-April 2017
  Proportion of mothers who report positive beliefs, self-efficacy, and perceptions of social norms about feeding animal source foods to children and feeding as often as usual during fasting based on questionnaire
Nutritional status of children 6-23 months of age | 2 years after baseline in a cross-sectional endline survey scheduled for March-April 2017
  Prevalence of stunting, underweight and wasting among children 6-23 months

CONTACTS AND LOCATIONS:
Overall Officials: Purnima Menon, PhD, Principal Investigator — International Food Policy Research Institute; Sunny S. Kim, PhD, Principal Investigator — International Food Policy Research Institute
Locations (1):
- International Food Policy Research Institute, Addis Ababa, Ethiopia

REFERENCES:
- [Derived] Kim SS, Nguyen PH, Tran LM, Alayon S, Menon P, Frongillo EA. Different Combinations of Behavior Change Interventions and Frequencies of Interpersonal Contacts Are Associated with Infant and Young Child Feeding Practices in Bangladesh, Ethiopia, and Vietnam. Curr Dev Nutr. 2019 Dec 9;4(2):nzz140. doi: 10.1093/cdn/nzz140. eCollection 2020 Feb. PMID 31976385
- [Derived] Kim SS, Nguyen PH, Yohannes Y, Abebe Y, Tharaney M, Drummond E, Frongillo EA, Ruel MT, Menon P. Behavior Change Interventions Delivered through Interpersonal Communication, Agricultural Activities, Community Mobilization, and Mass Media Increase Complementary Feeding Practices and Reduce Child Stunting in Ethiopia. J Nutr. 2019 Aug 1;149(8):1470-1481. doi: 10.1093/jn/nxz087. PMID 31165869
- See also: Alive & Thrive initiative website — http://aliveandthrive.org